CLINICAL TRIAL: NCT07005063
Title: Rotator Cuff Tendon Repair With FiberLocker System Patch Augmentation: A Prospective, Single-Arm, Non-Randomized, Pilot Study
Brief Title: Rotator Cuff Tendon Repair With FiberLocker System Patch Augmentation
Acronym: FIBERLOCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZuriMED Technologies AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZM072024; SNCTP000006378 (Other: Swiss National Trials Portal)
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Rotator Cuff Tear; Rotator Cuff Injury; Rotator Cuff Rupture
Keywords: Rotator cuff tear; Rotator cuff repair; Augmentation; Reinforcement; Mechanical augmentation
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augmentation of Rotator Cuff Repair using the FiberLocker System (Experimental): All enrolled participants will undergo repair of the rotator cuff tear, with augmentation utilizing the FiberLocker System.
  Interventions: Device: FiberLocker® System (encompassing SpeedPatch® PET and FiberLocker Instrument® SN)

INTERVENTIONS:
Device: FiberLocker® System (encompassing SpeedPatch® PET and FiberLocker Instrument® SN) — The FiberLocker® System is a mechanical augmentation system that includes an implant (SpeedPatch® PET) and an instrument (FiberLocker® Instrument SN) for its attachment. The implant is composed of non-woven PET fibers, and the instrument features a reciprocating needle at its tip, which pushes the individual patch fibers into the underlying tendon tissue

SUMMARY:
The overall objective of this clinical investigation is to assess the safety and efficacy of full-thickness arthroscopic rotator cuff repairs augmented with the FiberLocker System for the subjects. The primary outcome of the investigation is to assess the safety after full-thickness arthroscopic rotator cuff repairs augmented with the FiberLocker System in terms of postoperative adverse events through the 12-month follow-up. Main secondary outcomes include measures of efficacy and clinical performance evaluated at 6-week, 4.5-month, and 12-month follow-ups including retear rate assessed using MRI and different functional performance scores.

ELIGIBILITY:
Inclusion Criteria:

1. Subject requires surgical treatment of a full-thickness rotator cuff tear, according to Balgrist standard procedure
2. Full-thickness tear of the supraspinatus or combined infraspinatus and supraspinatus
3. The rotator cuff tear is of traumatic origin.
4. Subject is ≥ 40 years of age & ≤ 65 years of age.
5. Primary rotator cuff repair
6. Informed Consent signed by the subject
7. Pre-operative MRI performed

Exclusion Criteria:

1. Vulnerable subjects (as defined in ISO 14155)
2. Subjects who do not have the power of judgement or are unable to fully understand all aspects of the investigation that are relevant to the decision to participate
3. Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation,
4. Previous enrolment into the current investigation,
5. Enrolment of the PI, his/her family members, employees and other dependent persons,
6. Inability to follow the procedures of the investigation, or known or suspected non-compliance, e.g. due to language problems, psychological disorders, dementia, drug or alcohol abuse, etc. of the subject
7. Active smoker
8. History of claustrophobia that would prevent an MRI of the index shoulder
9. Presence of an implanted metallic device or other implants that would contraindicate acquisition or inhibit radiologist review of an MRI of the index shoulder
10. Pregnant or planning to become pregnant during the study period
11. Breast feeding women
12. Subject has conditions or circumstances that would interfere with study requirements.
13. Contraindications and limitations of the MD as described in the IFUs.
14. Partial rotator cuff tears
15. History or known allergy or intolerance to polyester
16. Complete full-thickness subscapularis tears greater than the superior 1/3 of the tendon, with Lafosse grade 3 or greater
17. Massive rotator cuff tears, tear size equal to or greater than 4 cm in the anterior-posterior dimension or irreparable rotator cuff tear
18. Limited space or exposure for implant delivery
19. Structural or pathological condition of the bone or soft tissue that could impair healing.
20. Intraoperative rotator cuff tear characteristics differ from preoperatively expected characteristics and fulfil one of the abovementioned criteria
21. Fatty infiltration of the index shoulder rotator cuff muscle > Goutallier Score 2
22. Corticosteroid injection in the operative shoulder within 6 weeks of operation
23. Subject shows frozen shoulder/adhesive capsulitis at day of surgery
24. Cases of moderate to severe osteoarthritis
25. Patients with inflammatory disease or auto-immune based joint diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, arthropathy)
26. Subjects with diabetes type I or II
27. The subject currently has an acute infection in the area surrounding the surgical site
28. Evidence of active infection, osteomyelitis, sepsis or distant infection which could spread to the index joint.
29. Any comorbidity or condition that renders the patient a poor surgical candidate as determined by the Investigator.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Total Number of Adverse Events (AEs) | Surgery to 12-month follow-up
  All operative and postoperative AEs will be recorded. Safety outcomes will be determined by evaluating the type, frequency, seriousness, and relationship to device or procedure of AEs for all subjects.
Total Number of Serious Adverse Events (SAEs) | Surgery to 12-month follow-up
  All operative and postoperative SAEs will be recorded. Safety outcomes will be determined by evaluating the type, frequency, and relationship to device or procedure of SAEs for all subjects.
Number of AE related to Device | Surgery to 12-month follow-up
  The operative and postoperative AEs that are related to the device will be reported. Safety outcomes will be determined by evaluating the type and frequency for all subjects.
Number of SAE related to Device | Surgery to 12-month follow-up
  The operative and postoperative SAEs that are related to the device will be reported. Safety outcomes will be determined by evaluating the type and frequency for all subjects.
Number of AE related to Procedure | Surgery to 12-month follow-up
  The operative and postoperative AEs that are related to the procedure will be reported. Safety outcomes will be determined by evaluating the type and frequency for all subjects.
Number of SAE related to Procedure | Surgery to 12-month follow-up
  The operative and postoperative SAEs that are related to the procedure will be reported. Safety outcomes will be determined by evaluating the type and frequency for all subjects.

SECONDARY OUTCOMES:
Retear Rate | 6-week, 4.5-month and 12-month follow-up
  Retears are defined as repairs showing structural defect of the tendon bone-interface on MRI according to type IV or V of the Sugaya classification. Cuff integrity according to the Sugaya classification is defined as follows: type I (repaired cuff of sufficientthickness, homogeneously low signal intensity), type II (sufficient thickness, partial high-signal intensity area), type III (insufficient thickness without discontinuity), type IV (minor discontinuity in 1 section, suggestive of a small tear), type V (major discontinuity in each image, suggestive of a medium-to-large tear).
Constant-Murley Score | Baseline and 12-month follow-up
  The Constant score will be calculated in a 100-point scale and compared with baseline. It will be measured with a patient-reported questionnaire & medical professional assessment at baseline and 12-month follow-up visit. A higher score indicates better function.
Visual Analog Scale for Pain (VAS) | Baseline, 2-week, 4.5-month and 12-month follow-up
  The VAS score will be calculated in a 0 to 10 scale and compared with baseline. Thereby, a higher score indicates greater pain intensity. VAS for average pain score over the last 24 hours will be assessed with a questionnaire.
Subjective Shoulder Value (SSV) Score | Baseline, 4.5-month and 12-month follow-up
  The SSV score is a patient-reported outcome measure used to assess a patient's perception of their shoulder function. It consists of a single question and each subject has to rate their shoulder function on a scale from 0% to 100%. Thereby, higher percentages indicates better shoulder function.
EQ-5D-5L survey | Baseline, 4.5-month and 12-month follow-up
  The EQ-5D-5L survey is a patient-reported outcome and consists of 2 parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system covers five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ VAS is the patient's self-rated health on a vertical visual analogue scale (0-100), whereas a higher score represents better health.
American Shoulder and Elbow Society (ASES) score | Baseline, 4.5-month and 12-month follow-up
  The ASES score is a patient-reported outcome measure survey which is completed by all subjects. It is used to assess shoulder function and pain. Based on the answers, a final score between 0 and 100 can be achieved. Thereby, higher scores indicate better shoulder function and less pain.
Sugaya Classification | 6-week, 4.5-month and 12-month follow-up
  The Sugaya Classification based on MRI images is used to evaluate the integrity of a repaired rotator cuff and to assess healing outcomes after a repair. The classification uses a categorial scoring system with grades from Type I to Type V.
  * Type I: repaired cuff of sufficient thickness, homogeneously low signal intensity
  * Type II: sufficient thickness, partial high-signal intensity area
  * Type III: insufficient thickness without discontinuity
  * Type IV: minor discontinuity in 1 section, suggestive of a small tear
  * Type V: major discontinuity in each image, suggestive of a medium-to-large tear
Goutallier Classification | Baseline, 6-week, 4.5-month and 12-month follow-up
  The Goutallier Classification is evaluated using MRI images to assess fatty infiltration and muscle degeneration in the rotator cuff. It has a categorial grading system from stage 0 to 4.
  Based on MRI images, the rotator cuff of each subject will be classified. Thereby, a higher classification means more fatty infiltration.
Tendon Thickness | Baseline, 6-week, 4.5-month and 12-month follow-up
  Tendon thickness of the affected rotator cuff tendon will be measured in a MRI images (in mm).
Fat Fraction of Muscle | Baseline, 6-week, 4.5-month and 12-month follow-up
  Fat fraction of muscle quantified in Dixon sequence will be evaluated on the MRI images. Accordingly, the range can be from 0% to 100%. A higher percentage indicates more fatty infiltration.

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided